CLINICAL TRIAL: NCT06480994
Title: Exclusion of Venous Thrombo-Embolism With a New Clinical Decision Support With Fresh Plasma, on Any Patient With VTE Suspicion
Brief Title: Exclusion of Venous Thrombo-Embolism With a New Clinical Decision Support
Acronym: EXTEND
Status: Recruiting | Type: Observational
Sponsor: Diagnostica Stago R&D (Industry)
Collaborators: Centre Hospitalier de Niort (Other); Centre Hospitalier le Mans (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: EXTEND 2021-A03135-36
Record Dates: First submitted 2024-06-17; First posted 2024-07-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism; Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Frozen plasma aliquots collected on citrated tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Routine Assays on fresh plasma — Routine coagulation tests using STA-R Max analyzer :
  Prothrombin Time (PT) activated Partial Thromboplastin Time (aPTT Thrombin Time (TT) Fibrinogen Anti-Xa activity
Diagnostic Test: New Clinical Decision Support on fresh plasma — D-Dimer and fibrin formation assays on STA-R Max analyzer. Calculation of the exclusion score using an algorithm (manual or based on Machine Learning) compared to a Clinical Decision Support cut-off.
Diagnostic Test: New Clinical Decision Support on frozen plasma — D-Dimer and fibrin formation assays on STA-R Max analyzer. Calculation of the exclusion score using an algorithm (manual or based on Machine Learning) compared to a Clinical Decision Support cut-off.

SUMMARY:
The goal of this non interventional study is to demonstrate the diagnostic performances on fresh plasmas in comparison with the performances on frozen plasmas in any patients with VTE suspicion, whatever the pre-test probability. The main question it aims to answer is :

Are the performances equivalent on fresh plasmas in comparison with frozen plasmas or is it necessary to determine a new algorithm of the Clinical Decision Support with a new cut-off? Participants will be diagnosed and treated in accordance with routine standard of care.

DETAILED DESCRIPTION:
Establish the diagnostic performance of the Clinical Decision Support tool on fresh plasma, in PE and in DVT, in comparison with that on frozen plasma, and in comparison with the current diagnostic strategy, on the entire population and on the following different subpopulations:

* Patients eligible for D-dimer assay, with low or moderate clinical probability, compared to the reference diagnosis (imaging and D-Dimer adjusted and not adjusted for age)
* Patients with high clinical probability, compared to the reference diagnosis (imaging)
* Patients not eligible for D-dimer assay: either with a condition associated with increased D-dimer levels in the absence of VTE, or with a history of PE or DVT for less than 3 months or suspected thrombotic events
* Patients with known and active cancer
* Patients with COVID-19. The assays will be conducted on a fresh and frozen plasma aliquots.

ELIGIBILITY:
Inclusion Criteria:

* PE and/or DVT suspicion
* No opposition after informing the patient for his participation in research and processing of their data for this purpose,
* Benefiting from the social security system

Exclusion Criteria:

* Preventive or curative anticoagulant treatment, or fibrinolytic treatment,
* Legal protection (e.g. guardianship or curatorship),
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients eligible for D-dimer assay, with low or moderate clinical probability, compared to the reference diagnosis (imaging and D-Dimer adjusted and not adjusted for age)
  * Patients with high clinical probability, compared to the reference diagnosis (imaging)
  * Patients not eligible for D-dimer assay: either with a condition associated with increased D-dimer levels in the absence of VTE, or with a history of PE or DVT for less than 3 months or suspected thrombotic events
  * Patients with known and active cancer
  * Patients with COVID-19
Sampling Method: Probability Sample
Enrollment: 1836 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of the new clinical decision support with fresh plasma | 37 months
  Reproducibility (%) calculated with 70% of the study population with fresh plasma in comparison with frozen plasma.
Threshold of the new clinical decision support with fresh plasma | 37 months
  Threshold calculated with 70% of the study population with fresh plasma in comparison with frozen plasma.
PE / DVT sensitivity of the clinical decision support | 48 months
  Sensitivity of the clinical decision support with fresh plasma in comparison with reference diagnosis.
PE / DVT specificity of the clinical decision support | 48 months
  Specificity of the clinical decision support with fresh plasma in comparison with reference diagnosis.
PE / DVT likelihood ratio of the clinical decision support | 48 months
  Likelihood ratio of the clinical decision support with fresh plasma in comparison with reference diagnosis.
PE / DVT exclusion percentage of the clinical decision support | 48 months
  Exclusion percentage of the clinical decision support with fresh plasma in comparison with reference diagnosis.
PE / DVT negative predictive value of the clinical decision support | 48 months
  Negative Predictive Value of the clinical decision support with fresh plasma in comparison with reference diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT VIOLEAU, Principal Investigator — Centre Hospitalier de Niort
Locations (4):
- France (4):
  - Centre Hospitalier de Niort, Niort, Sartres
  - Centre Hospitalier le Mans, Le Mans, Sartre
  - CHU Dijon Bourgogne, Dijon
  - University Hospital Grenoble, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Contant G., Mirshahi S.S., Depasse F., Soria J. A new D-dimer concept for more specific detection of venous thromboembolism. Res Pract Thromb Haemost 2017; 1, (Suppl. 1), PB 1385, Abstracts of the XXVI Congress of the International Society on Thrombosis and Haemostasis, July 8-13, 2017
- [Background] Planquette B, Jumel S, Pastre J, Pereira H, Marey J, Roche A, Chatellier G, Sanchez O and Meyer G. SOFIE: Soluble Fibrin for Diagnosing Pulmonary Embolism. Res Pract Thromb Haemost 2017; 1, (Suppl. 1), PB 1393, Abstracts of the XXVI Congress of the International Society on Thrombosis and Haemostasis, July 8-13, 2017.
- [Background] Heit JA, Cohen AT, Anderson FA. Estimated annual number of incident and recurrent, non-fatal and fatal venous thromboembolism (VTE) events in the US. Blood 2005;106(11):910
- [Background] Cohen AT, Agnelli G, Anderson FA, Arcelus JI, Bergqvist D, Brecht JG, Greer IA, Heit JA, Hutchinson JL, Kakkar AK, Mottier D, Oger E, Samama MM, Spannagl M; VTE Impact Assessment Group in Europe (VITAE). Venous thromboembolism (VTE) in Europe. The number of VTE events and associated morbidity and mortality. Thromb Haemost. 2007 Oct;98(4):756-64. doi: 10.1160/TH07-03-0212. PMID 17938798
- [Background] ISTH Steering Committee for World Thrombosis Day. Thrombosis: a major contributor to the global disease burden. J Thromb Haemost. 2014 Oct;12(10):1580-90. doi: 10.1111/jth.12698. PMID 25302663
- [Background] Anderson FA Jr, Spencer FA. Risk factors for venous thromboembolism. Circulation. 2003 Jun 17;107(23 Suppl 1):I9-16. doi: 10.1161/01.CIR.0000078469.07362.E6. PMID 12814980
- [Background] Wells PS. Integrated strategies for the diagnosis of venous thromboembolism. J Thromb Haemost. 2007 Jul;5 Suppl 1:41-50. doi: 10.1111/j.1538-7836.2007.02493.x. PMID 17635707
- [Background] Wells PS, Anderson DR, Bormanis J, Guy F, Mitchell M, Gray L, Clement C, Robinson KS, Lewandowski B. Value of assessment of pretest probability of deep-vein thrombosis in clinical management. Lancet. 1997 Dec 20-27;350(9094):1795-8. doi: 10.1016/S0140-6736(97)08140-3. PMID 9428249
- [Background] Le Gal G, Righini M, Roy PM, Sanchez O, Aujesky D, Bounameaux H, Perrier A. Prediction of pulmonary embolism in the emergency department: the revised Geneva score. Ann Intern Med. 2006 Feb 7;144(3):165-71. doi: 10.7326/0003-4819-144-3-200602070-00004. PMID 16461960
- [Background] Schulman S, Ageno W, Konstantinides SV. Venous thromboembolism: Past, present and future. Thromb Haemost. 2017 Jun 28;117(7):1219-1229. doi: 10.1160/TH16-10-0823. Epub 2017 Jun 8. PMID 28594049
- [Background] Di Nisio M, Squizzato A, Rutjes AW, Buller HR, Zwinderman AH, Bossuyt PM. Diagnostic accuracy of D-dimer test for exclusion of venous thromboembolism: a systematic review. J Thromb Haemost. 2007 Feb;5(2):296-304. doi: 10.1111/j.1538-7836.2007.02328.x. Epub 2006 Nov 28. PMID 17155963
- [Background] Righini M. Is it worth diagnosing and treating distal deep vein thrombosis? No. J Thromb Haemost. 2007 Jul;5 Suppl 1:55-9. doi: 10.1111/j.1538-7836.2007.02468.x. PMID 17635709
- [Background] Pawelec G, Goldeck D, Derhovanessian E. Inflammation, ageing and chronic disease. Curr Opin Immunol. 2014 Aug;29:23-8. doi: 10.1016/j.coi.2014.03.007. Epub 2014 Apr 22. PMID 24762450
- [Background] Tita-Nwa F, Bos A, Adjei A, Ershler WB, Longo DL, Ferrucci L. Correlates of D-dimer in older persons. Aging Clin Exp Res. 2010 Feb;22(1):20-3. doi: 10.1007/BF03324810. PMID 20305364
- [Background] Harper PL, Theakston E, Ahmed J, Ockelford P. D-dimer concentration increases with age reducing the clinical value of the D-dimer assay in the elderly. Intern Med J. 2007 Sep;37(9):607-13. doi: 10.1111/j.1445-5994.2007.01388.x. Epub 2007 Jun 2. PMID 17543005
- [Background] Righini M, Le Gal G, Bounameaux H. Venous thromboembolism diagnosis: unresolved issues. Thromb Haemost. 2015 Jun;113(6):1184-92. doi: 10.1160/TH14-06-0530. Epub 2014 Dec 11. PMID 25503584
- [Background] Huisman MV, Klok FA. Current challenges in diagnostic imaging of venous thromboembolism. Blood. 2015 Nov 19;126(21):2376-82. doi: 10.1182/blood-2015-05-640979. PMID 26585807
- [Background] Righini M, Le Gal G, Perrier A, Bounameaux H. The challenge of diagnosing pulmonary embolism in elderly patients: influence of age on commonly used diagnostic tests and strategies. J Am Geriatr Soc. 2005 Jun;53(6):1039-45. doi: 10.1111/j.1532-5415.2005.53309.x. PMID 15935031
- [Background] van Belle A, Buller HR, Huisman MV, Huisman PM, Kaasjager K, Kamphuisen PW, Kramer MH, Kruip MJ, Kwakkel-van Erp JM, Leebeek FW, Nijkeuter M, Prins MH, Sohne M, Tick LW; Christopher Study Investigators. Effectiveness of managing suspected pulmonary embolism using an algorithm combining clinical probability, D-dimer testing, and computed tomography. JAMA. 2006 Jan 11;295(2):172-9. doi: 10.1001/jama.295.2.172. PMID 16403929
- [Background] Pernod G, Caterino J, Maignan M, Tissier C, Kassis J, Lazarchick J; DIET study group. D-Dimer Use and Pulmonary Embolism Diagnosis in Emergency Units: Why Is There Such a Difference in Pulmonary Embolism Prevalence between the United States of America and Countries Outside USA? PLoS One. 2017 Jan 13;12(1):e0169268. doi: 10.1371/journal.pone.0169268. eCollection 2017. PMID 28085911
- [Background] Righini M, Van Es J, Den Exter PL, Roy PM, Verschuren F, Ghuysen A, Rutschmann OT, Sanchez O, Jaffrelot M, Trinh-Duc A, Le Gall C, Moustafa F, Principe A, Van Houten AA, Ten Wolde M, Douma RA, Hazelaar G, Erkens PM, Van Kralingen KW, Grootenboers MJ, Durian MF, Cheung YW, Meyer G, Bounameaux H, Huisman MV, Kamphuisen PW, Le Gal G. Age-adjusted D-dimer cutoff levels to rule out pulmonary embolism: the ADJUST-PE study. JAMA. 2014 Mar 19;311(11):1117-24. doi: 10.1001/jama.2014.2135. PMID 24643601
- [Background] van der Hulle T, Cheung WY, Kooij S, Beenen LFM, van Bemmel T, van Es J, Faber LM, Hazelaar GM, Heringhaus C, Hofstee H, Hovens MMC, Kaasjager KAH, van Klink RCJ, Kruip MJHA, Loeffen RF, Mairuhu ATA, Middeldorp S, Nijkeuter M, van der Pol LM, Schol-Gelok S, Ten Wolde M, Klok FA, Huisman MV; YEARS study group. Simplified diagnostic management of suspected pulmonary embolism (the YEARS study): a prospective, multicentre, cohort study. Lancet. 2017 Jul 15;390(10091):289-297. doi: 10.1016/S0140-6736(17)30885-1. Epub 2017 May 23. PMID 28549662
- [Background] Freund Y, Cachanado M, Aubry A, Orsini C, Raynal PA, Feral-Pierssens AL, Charpentier S, Dumas F, Baarir N, Truchot J, Desmettre T, Tazarourte K, Beaune S, Leleu A, Khellaf M, Wargon M, Bloom B, Rousseau A, Simon T, Riou B; PROPER Investigator Group. Effect of the Pulmonary Embolism Rule-Out Criteria on Subsequent Thromboembolic Events Among Low-Risk Emergency Department Patients: The PROPER Randomized Clinical Trial. JAMA. 2018 Feb 13;319(6):559-566. doi: 10.1001/jama.2017.21904. PMID 29450523
- [Background] Penaloza A, Soulie C, Moumneh T, Delmez Q, Ghuysen A, El Kouri D, Brice C, Marjanovic NS, Bouget J, Moustafa F, Trinh-Duc A, Le Gall C, Imsaad L, Chretien JM, Gable B, Girard P, Sanchez O, Schmidt J, Le Gal G, Meyer G, Delvau N, Roy PM. Pulmonary embolism rule-out criteria (PERC) rule in European patients with low implicit clinical probability (PERCEPIC): a multicentre, prospective, observational study. Lancet Haematol. 2017 Dec;4(12):e615-e621. doi: 10.1016/S2352-3026(17)30210-7. Epub 2017 Nov 14. PMID 29150390
- [Background] Wolberg AS. Thrombin generation and fibrin clot structure. Blood Rev. 2007 May;21(3):131-42. doi: 10.1016/j.blre.2006.11.001. Epub 2007 Jan 8. PMID 17208341
- [Background] Undas A. Prothrombotic Fibrin Clot Phenotype in Patients with Deep Vein Thrombosis and Pulmonary Embolism: A New Risk Factor for Recurrence. Biomed Res Int. 2017;2017:8196256. doi: 10.1155/2017/8196256. Epub 2017 Jun 27. PMID 28740853
- [Background] Zabczyk M, Undas A. Plasma fibrin clot structure and thromboembolism: clinical implications. Pol Arch Intern Med. 2017 Dec 22;127(12):873-881. doi: 10.20452/pamw.4165. Epub 2017 Dec 11. PMID 29225327
- [Background] Undas A. How to Assess Fibrinogen Levels and Fibrin Clot Properties in Clinical Practice? Semin Thromb Hemost. 2016 Jun;42(4):381-8. doi: 10.1055/s-0036-1579636. Epub 2016 Apr 12. PMID 27071050
- [Background] Schafer M, Werner S. Cancer as an overhealing wound: an old hypothesis revisited. Nat Rev Mol Cell Biol. 2008 Aug;9(8):628-38. doi: 10.1038/nrm2455. Epub 2008 Jul 16. PMID 18628784
- [Background] Thachil J, Tang N, Gando S, Falanga A, Cattaneo M, Levi M, Clark C, Iba T. ISTH interim guidance on recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 May;18(5):1023-1026. doi: 10.1111/jth.14810. Epub 2020 Apr 27. No abstract available. PMID 32338827
- [Background] Mahé I, Chidiac J, Djennaoui S, Javaud N, Planquette B, Peynaud-Debayle E, Sofiane Baccar L, Dumont B, Meyer G, Contant G, Depasse F, Siguret V, Helfer H. Evaluation of the Fibrin Assay for Venous Thromboembolism Exclusion in Cancer Patients: Subanalysis of a Prospective Assessment (FSET STUDY). Blood 134(Supplement_1):3663-3663, November 2019